CLINICAL TRIAL: NCT04393246
Title: mulTi-Arm Therapeutic Study in Pre-ICu Patients Admitted With Covid-19 - Experimental Drugs and Mechanisms (TACTIC-E)
Brief Title: mulTi-Arm Therapeutic Study in Pre-ICu Patients Admitted With Covid-19 - Experimental Drugs and Mechanisms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Joseph Cheriyan, MD, Consultant in Clinical Pharmacology, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TACTIC-E
Record Dates: First submitted 2020-05-16; First posted 2020-05-19 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — dapagliflozin; ambrisentan; Standard of Care

STUDY DESIGN:
Intervention Model Description: TACTIC-E is a randomised, parallel arm, open-label platform trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of care (Active Comparator): Standard of care
  Interventions: Other: Standard of care
- EDP1815 (Experimental): 1.6 x 10^11 cells dosage-in-capsule orally twice per day for up to 7 days (with the option to extend up to 14 days), on top of standard of care
  Interventions: Drug: EDP1815
- Dapagliflozin and Ambrisentan (Experimental): Ambrisentan 5mg tablet orally once per day for up to a maximum of 14 days and Dapagliflozin 10mg tablet orally once per day for up to a maximum of 14 days, on top of standard of care
  Interventions: Drug: Dapagliflozin; Drug: Ambrisentan

INTERVENTIONS:
Drug: EDP1815 — EDP1815 is an orally administered pharmaceutical preparation of a single strain of Prevotella histicola isolated from the duodenum of a human donor. EDP1815 is currently in phase 2 clinical development and has European and US approval to initiate a multinational psoriasis study.
  Arms: EDP1815
Drug: Dapagliflozin — Dapagliflozin is a sodium-glucose co-transporter 2 (SGLT-2) inhibitor. Dapagliflozin is licensed for use in the UK for treatment of Type II diabetes. Since this trial is evaluating Dapagliflozin in an unlicensed indication, it is being carried out under a Clinical Trial Authorisation (CTA)
  Other Names: Forxiga
  Arms: Dapagliflozin and Ambrisentan
Drug: Ambrisentan — Ambrisentan is an endothelin receptor antagonist, and is selective for the type A endothelin receptor (ETA). Ambrisentan was approved by the U.S. Food and Drug Administration (FDA) and the European Medicines Agency (EMA) and indicated for the treatment of pulmonary arterial hypertension.
  Other Names: Letairis, Volibris, Pulmonext
  Arms: Dapagliflozin and Ambrisentan
Other: Standard of care — Regular standard of care for COVID-19 patients
  Arms: Standard of care

SUMMARY:
TACTIC-E is a randomised, parallel arm, open-label platform trial for investigating potential treatments for COVID-19 disease. While SARS-CoV infection evades detection by the immune system in the first 24 hours of infection, it ultimately produces a massive immune system response in the subgroup of people who develop severe complications. Most tissue damage following infection with COVID-19 appears to be due to a later, exaggerated, host immune response (Gralinski and Baric 2015). This leads to lung and sometimes multi-organ damage.

Most people who develop these severe complications still have virus present in their respiratory tract at the time-point when the disease starts to evolve. Immune modulation in the presence of active infection has potential to cause more harm than benefit. Safety considerations when studying immune modulation strategies are paramount. This study will assess the efficacy of a novel immunomodulatory agent and a novel combination of approved agents which may protect the patient against end-organ damage and modulate the pulmonary vascular response. This study will compare the novel therapeutic agent EDP1815 and a novel combination of the approved agents dapagliflozin and ambrisentan against Standard of Care. A trial arm (UNI911) with the IMP Niclosamide was added to the protocol with one patient recruited into this arm. Following an AESI and after discussions between the funder and the Sponsor the arm was stopped.

DETAILED DESCRIPTION:
TACTIC-E will assess the efficacy of the novel immunomodulatory agent EDP1815 and a combination of the approved cardiovascular drugs dapagliflozin and ambrisentan as potential treatments for COVID-19 disease against Standard of Care alone. These agents target the dysregulated immune response that drive the severe lung, and other organ, damage frequently seen during COVID-19 infection, with an aim to promote a positive vascular response to reduce end-organ damage.

Treatment with EDP1815 will be for up to 7 days, with the option of extension to 14 days at the discretion of the PI or their delegate, if the patient is felt to be clinically responding to treatment, is tolerating treatment, and is judged to be likely to benefit from a longer treatment course. Treatment with combination dapagliflozin and ambrisentan will be for up to 14 days. Patients will be randomised in a 1:1:1 ratio across treatments.

TACTIC-E will use a platform design with interim analysis to make efficient decisions about efficacy and futility (e.g. lack of efficacy and risk of harm) of the trial treatments. This enables the trial to stop recruiting to arms early where a clear efficacy decision can be made. It also allows for the addition of further arms.

ELIGIBILITY:
General Inclusion Criteria:

* Be aged 18 and over
* Have clinical picture strongly suggestive of COVID-19-related disease (with/without positive COVID-19 test) AND

  * Risk count (as defined below) >3 OR
  * Risk count ≥3 if it includes "Radiographic severity score >3"
* Be hospitalized or eligible for hospitalization on clinical grounds
* Be considered an appropriate subject for intervention with immunomodulatory or other disease modifying agents in the opinion of the investigator
* Is able to swallow capsules/tablets

General Exclusion Criteria:

* Inability to supply direct informed consent from patient or from Next of Kin or Independent Healthcare Provider on behalf of patient
* Invasive mechanical ventilation at time of screening
* Contraindications to study drugs, including hypersensitivity to the active substances or any of the excipients
* Currently on any of the study investigational medicinal products
* Concurrent participation in an interventional clinical trial (observational studies allowed)
* Patient moribund at presentation or screening
* Pregnancy at screening
* Unwilling to stop breastfeeding during treatment period
* Known severe hepatic impairment (with or without cirrhosis)
* Requiring dialysis Cockcroft Gault estimated creatinine clearance < 30 ml /min/1.73m2 at screening
* Inability to swallow at screening visit
* Any medical history or clinically relevant abnormality that is deemed by the principal investigator and/or medical monitor to make the patient ineligible for inclusion because of a safety concern.

EDP1815-Specific Exclusion Criteria:

* Patient is taking a systemic immunosuppressive agent such as, but not limited to, oral steroids, methotrexate, azathioprine, ciclosporin or tacrolimus, unless these are given as part of COVID standard of care treatment.
* Patient has known primary or secondary B cell disorder

Dapagliflozin- and Ambrisentan-Specific Exclusion Criteria:

* Type 1 diabetes
* Known idiopathic pulmonary fibrosis
* Previous hospital admission with ketoacidosis
* Patients concurrently on other SGLT2 inhibitors
* History of symptomatic heart failure within 3 months of admission
* Sustained blood pressure below 100/70 mmHg at admission
* Metabolic acidosis defined as pH< 7.25 AND ketones > 3.0 mmol/L
* Alanine transaminase and/or aspartate transaminase (ALT and/or AST) > 3 times the upper limit of normal (only one needs to be measured)

Risk Count

Patients will be given a Risk Count equal to the cumulative points received for the following criteria (no = 0 points, yes = 1 point):

Male gender, Age > 40 years, Non-white ethnicity, Diabetes, Hypertension, Neutrophils > 8.0x10^9/L, CRP > 40mg/L, Radiographic severity score >3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Time to incidence of the composite endpoint of: Death, Mechanical ventilation, ECMO, Cardiovascular organ support, or Renal failure | up to Day 14
  Number of days taken for occurrence of one of the following events: 1. Death 2. Mechanical ventilation 3. Extracorporeal membrane oxygenation (ECMO) 4. Cardiovascular organ support (balloon pump or inotropes/vassopressors) 5. Renal failure (estimated creatinine clearance (by Cockcroft-Gault formula) <15 ml /min/1.73m^2), haemofiltration or dialysis

SECONDARY OUTCOMES:
Change in biomarkers thought to be associated with progression of COVID-19 compared to baseline: IL-6 | 14 days
  Change in patient blood levels of IL-6 compared to baseline, measured in pg/mL
Change in biomarkers thought to be associated with progression of COVID-19 compared to baseline: ferritin | 14 days
  Change in patient blood levels of ferritin compared to baseline, measured in ng/mL
Change in biomarkers thought to be associated with progression of COVID-19 compared to baseline: c-reactive protein (CRP) | 14 days
  Change in patient blood levels of CRP compared to baseline, measured in mg/L
Change in biomarkers thought to be associated with progression of COVID-19 compared to baseline: D-dimer | 14 days
  Change in patient blood levels of D-dimer compared to baseline, measured in ng/mL
Change in biomarkers thought to be associated with progression of COVID-19 compared to baseline: neutrophil/lymphocyte ratio | 14 days
  Change in patient blood levels of neutrophil/lymphocyte ratio compared to baseline
Change in biomarkers thought to be associated with progression of COVID-19 compared to baseline: lactate dehydrogenase (LDH) | 14 days
  Change in patient blood levels of lactate dehydrogenase (LDH) compared to baseline, measured in U/L
Change in clinical status as assessed on 7-point ordinal scale compared to baseline | 14 days
  The clinical status of the patients is assessed using 7-point ordinal scale as follows: 1 = Death, 2 = Mechanical ventilation, 3 = Non-invasive or high flow oxygen, 4 = Low flow oxygen, 5 = Hospitalised - no oxygen, 6 = Discharged - normal activities not resumed, 7 = Discharged - normal activities resumed
Time to each of the individual endpoints of the composite primary outcome measure | 14 days
  Number of days taken for occurrence of each of the following events: 1. Death 2. Mechanical ventilation 3. Extracorporeal membrane oxygenation (ECMO) 4. Cardiovascular organ support (balloon pump or inotropes/vassopressors) 5. Renal failure (estimated creatinine clearance (by Cockcroft-Gault formula) <15 ml /min/1.73m^2), haemofiltration or dialysis
Proportion of patients with adverse events of special interest in each treatment arm | 14 days
  The proportion of patients in each treatment arm that experience adverse events of special interest, defined as: Diabetic ketoacidosis in patients on Ambrisentan & Dapagliflozin, New peripheral oedema in patients on Ambrisentan & Dapagliflozin arm
Time to Sp02 >94% on room air | 14 days
  The time taken to achieve blood oxygen saturation levels above 94% in patients on room air, measured in hours/days (chronically hypoxic individuals will be excluded from this analysis)
Time to first negative SARS-CoV2 PCR | 14 days
  The amount of time between a patient's first positive SARS-CoV2 PCR test and a patient's first negative SARS-CoV2 PCR test, measured in days
Duration of oxygen therapy | 14 days
  The duration of oxygen therapy given to a patient, measured in days
Duration of hospitalisation | 14 days
  The duration of hospitalisation of a patient, measured in days
All-cause mortality at day 28 | 28 days
  The number of deaths recorded at 28 days irrespective of the cause
Time to clinical improvement | 14 days
  The time to clinical improvement for a patient, defined as: >2 point improvement from Day 1 on the 7-point ordinal scale, measured in days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MBChB MA FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gralinski LE, Baric RS. Molecular pathology of emerging coronavirus infections. J Pathol. 2015 Jan;235(2):185-95. doi: 10.1002/path.4454. PMID 25270030
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Lu IN, Kulkarni S, Fisk M, Kostapanos M, Banham-Hall E, Kadyan S, Bond S, Norton S, Cope A, Galloway J, Hall F, Jayne D, Wilkinson IB, Cheriyan J. muLTi-Arm Therapeutic study in pre-ICu patients admitted with Covid-19-Experimental drugs and mechanisms (TACTIC-E): A structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Jul 31;21(1):690. doi: 10.1186/s13063-020-04618-2. PMID 32736592